CLINICAL TRIAL: NCT03635008
Title: Effects of Anodal Transcranial Direct Current Stimulation Over the Contralesional Hemisphere on Motor Recovery in Subacute Stroke Patients With Severe Upper Extremity Hemiparesis: Study Protocol for a Randomized Controlled Trial
Brief Title: Anodal Transcranial Direct Current Stimulation Over the Contralesional Hemisphere on Motor Recovery in Subacute Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: the Ministry of Trade, Industry & Energy(MOTIE, Korea), Ybrain (Korea) (Unknown)
Responsible Party: Principal Investigator, Won-Seok Kim, Assistant Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-1805/468-002
Record Dates: First submitted 2018-07-14; First posted 2018-08-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Stroke; Transcranial Direct Current Stimulation; Recovery of Function; Neurological Rehabilitation
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, sham-controlled, parallel group design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An investigator who applies the tDCS to the participants will not be masked. However, other investigators including outcome assessors and participants will be masked. The other care providers in our department (e.g. other physio- or occupational therapists) will be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS (Experimental): This group will receive the 25 mins of the tDCS (Yrain, Korea) over the contralesional premotor area simultaneously with 25 mins of the robotic arm training using Armeo Power (Hocoma, Switzerland), per day. Additional 30 mins of occupational therapy focusing on the arm motor recovery will be provided per day. These interventions will be provided for 10 weekdays. Other conventional rehabilitation (e.g. gait training, speech therapy) will be permitted.
  Regard to the anodal tDCS, the anode will be placed over the contralesional premotor area (2.5 cm anterior to the C3 or C4 in 10-20 EEG system) and cathode will be placed over the contralateral supraorbital area. The stimulation intensity will be 2mA.
  Interventions: Device: tDCS
- sham tDCS (Placebo Comparator): This group will receive the 25 mins of the tDCS (Yrain, Korea) over the contralesional premotor area simultaneously with 25 mins of the robotic arm training using Armeo Power (Hocoma, Switzerland), per day. Additional 30 mins of occupational therapy focusing on the arm motor recovery will be provided per day. These interventions will be provided for 10 weekdays. Other conventional rehabilitation (e.g. gait training, speech therapy) will be permitted.
  Regard to the sham tDCS, the anode will be placed over the contralesional premotor area (2.5 cm anterior to the C3 or C4 in 10-20 EEG system) and cathode will be placed over the contralateral supraorbital area. The stimulation intensity will be started but the intensity will decrease and stop in 30 seconds.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Regard to the anodal tDCS, the anode will be placed over the contralesional premotor area (2.5 cm anterior to the C3 or C4 in 10-20 EEG system) and cathode will be placed over the contralateral supraorbital area. The stimulation intensity will be 2mA. For the sham tDCS the stimulation will be applied for just first 30 seconds.

SUMMARY:
Upper limb recovery is not predicted by the initial severity of paralysis and the parameters reflecting the integrity of the corticospinal tract (e.g. motor evoked potential, fractional anisotropy in diffusion tensor imaging). Although the inhibition of the contralesional hemisphere is known to be beneficial for the upper limb recovery after stroke in previous studies, this is not proven in the severely paralyzed upper limb. And the studies using the noninvasive stimulation in subacute stroke is lack. In addition, the role of contralesional (unaffected) hemisphere is known to be playing the important role in severe stroke.

In this randomized, double-blind, sham-controlled studies, the patients with subacute stroke (<3 months after stroke onset), severe paralysis of the upper limb with poor prognosis (poor motor score and no response of motor evoked potential recorded in the extensor carpi radialis muscle) will be recruited. Interventional group will receive the 25 mins of anodal transcranial direct current stimulation (tDCS) over the contralesional premotor area plus 25 mins of robotic arm training per session for 10 sessions in 2 weeks. Control group will receive the same treatment except for sham tDCS instead of anodal tDCS over the contralesional premotor area. Functional outcome will be measured before and after the intervention (baseline, immediately after the intervention and 1 month after the intervention). Cortical activation pattern will be measured by the electroencephalography (EEG) at baseline and immediately after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-85 years old
* Ischemic or Hemorrhagic stroke confirmed by the MRI or CT
* First-ever stroke
* < 3 months after stroke
* Unilateral upper limb weakness due to the stroke and meets the following all conditions: (1)Shoulder Abduction Finger Extension (SAFE) score (range 0-10) revealing the motor paralysis is below 8 (lower score mean worse function)), (2)Fugl Meyer Assessment score in the affected upper extremity is 25 or under 25. (3)No response in the motor evoked potential recorded on the affected extensor carpi radialis muscle,

Exclusion Criteria:

* recurrent stroke
* history of the other brain injury (e.g. traumatic brain injury)
* poor cognitive function (score of korean version of mini-mental state exam is 15 or below 15).
* Poor cooperation due to delirium or problems in the consciousness
* Uncontrolled or unstable medical conditions.
* Pregnant
* Scalp problems which interfere with the tDCS application
* Robotic arm training can not be applied due to the unstable sitting posture or head control, or arm pain.
* Metals in the head (e.g. clip, coil)
* Cardiac pacemaker or cochlear implants

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) scores of the upper extremity | Change from Baseline FMA at 2 weeks
  range: 0 (worst) -66 (best)

SECONDARY OUTCOMES:
Korean version of modified Barthel Index (K-MBI) | Change from baseline K-MBI at 2 weeks
  range: 0 (worst) -100 (best)
Korean version of modified Barthel Index (K-MBI) | Change from baseline K-MBI at 6 weeks
  range: 0 (worst) -100 (best)
Brunnstrom stage (B-stage) of arm | Change from baseline B-stage at 2 weeks
  range: 1(worst) -6 (best)
Brunnstrom stage (B-stage) of arm | Change from baseline B-stage at 6 weeks
  range: 1(worst) -6 (best)
Box and Block Test (BBT) | Change from baseline BBT at 2 weeks
  maximum number of blocks from one compartment of a box to another of equal size, within 60 seconds, more numbers mean better function
Box and Block Test (BBT) | Change from baseline BBT at 6 weeks
  maximum number of blocks from one compartment of a box to another of equal size, within 60 seconds, more numbers mean better function
Modified Ashworth Scale | 2 weeks after baseline
  to measure the spasticity: 6 grades: 0 (no spasticity), 1, 1+, 2, 3, 4 (severe spasticity)
Modified Ashworth Scale | 6 weeks after baseline
  to measure the spasticity: 6 grades: 0 (no spasticity), 1, 1+, 2, 3, 4 (severe spasticity)
Manual muscle power test | 2 weeks after baseline
  3 proximal (shoulder abduction, elbow flexion, and extension) and 5 distal (flexion and extension of the hand and fingers, and thumb flexion) muscle groups, 6 grades ranges from 0 (flaccid) to 5 (strongest).
Manual muscle power test | 6 weeks after baseline
  3 proximal (shoulder abduction, elbow flexion, and extension) and 5 distal (flexion and extension of the hand and fingers, and thumb flexion) muscle groups, 6 grades ranges from 0 (flaccid) to 5 (strongest).
Laterality Index | 2 weeks after baseline
  Ratio of the cortical activation between the contra- and ipsilesional motor area recorded by the electroencephalography
Laterality Index | 6 weeks after baseline
  Ratio of the cortical activation between the contra- and ipsilesional motor area recorded by the electroencephalography
Fugl-Meyer Assessment (FMA) scores of the upper extremity | Change from Baseline FMA at 6 weeks
  range: 0 (worst) -66 (best)

CONTACTS AND LOCATIONS:
Overall Officials: Won-Seok Kim, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Please Select, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
We are not planning to share the individual data publicly. However, if other researchers interested in our project, they can contact PI by email and we can discuss further for the sharing. If data sharing is decided after the discussion with other researchers, we will consider sharing after the review of the appropriateness by our institutional review board.